CLINICAL TRIAL: NCT03279172
Title: A Comparison of Videolaryngoscope and Direct Laryngoscope in Intraocular Pressure Changes, Throat Pain, Intubation Time and Hemodynamic Variables
Brief Title: A Comparison of Videolaryngoscope and Direct Laryngoscope in IOP Changes, Throat Pain, IT and Hemodynamic Variables
Acronym: IOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Ceyda Ozhan Caparlar, Principle investigator, Clinical Specialist of anesthesiology, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22051012
Record Dates: First submitted 2017-08-07; First posted 2017-09-12 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Intraocular Pressure; Intubation;Difficult
Keywords: videolaryngoscope; intraocular pressure; Direct laryngoscope

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Direct Laryngoscope (Experimental): direct laryngoscope (macintosh laryngoscope) is used in elective surgeries with maximal duration time for two hours. Standard anaesthesia was used on group and BIS monitorisation was applied. A record was made of IOP, hemodynamic changes and oxygen saturation at 3 and 10 minutes after intubation. Throat pain was evaluated by questioning the patient at 10 minutes and 24 hours after waking from general anaesthesia. The duration of intubation was recorded as the time from the laryngoscope entering the mouth to removal with end-tidal carbon dioxide on the monitor. Macintosh laryingoscope, BIS monitoring and tonometry would be used in Group Direct Laryngoscope.
  Interventions: Procedure: direct laryngoscope; Procedure: videolaryngoscope
- Group videolaryngoscope (Experimental): Videolaryngoscope is used in elective surgeries with maximal duration time for two hours. Standard anaesthesia was used on group and BIS monitorisation was applied. A record was made of IOP, hemodynamic changes and oxygen saturation at 3 and 10 minutes after intubation. Throat pain was evaluated by questioning the patient at 10 minutes and 24 hours after waking from general anaesthesia. The duration of intubation was recorded as the time from the laryngoscope entering the mouth to removal with end-tidal carbon dioxide on the monitor. Video laryingoscope, BIS monitoring and tonometry would be used in Group Video Laryngoscope.
  Interventions: Procedure: direct laryngoscope; Procedure: videolaryngoscope

INTERVENTIONS:
Procedure: direct laryngoscope — procedure entubatıon
Procedure: videolaryngoscope

SUMMARY:
The aim of the study was to compare intraocular pressure, intubation time, throat pain and hemodynamic variables using direct or videolaryngoscopy under general anesthesia requiring endotracheal intubation

DETAILED DESCRIPTION:
INTRODUCTION Videolaryngoscopes are the new generation devices which were introduced into the difficult intubation algorithm by the American Society of Anaesthesiologists (ASA) in 2013 (1). Videolaryngoscopes are known to be superior to traditional direct laryngoscopy in cases of difficult airway, glottic visualisation is obtained more easily and less airway trauma is seen (2). Portable videolaryngoscope which is used in difficult airways (3). There are 2, 3, and 4 numbered blades. In the light source of the blade of the videolaryngoscope, there is a camera which is connected to a video screen monitor. In addition to passing soft tissues by visualisation, the camera is helpful in defining the glottic appearance (1).

There are studies which have compared the hemodynamic response and increase in IOP in intubation using direct laryngoscope and various videolaryngoscopes and airway devices . However, to the best of our knowledge there is no study comparing the effect on the increase in IOP of videolaryngoscope and direct laryngoscope. The aim of the current study was to compare IOP, hemodynamic parameters and throat pain in the use of videolaryngoscope and the direct laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgery under general anaesthesia

Exclusion Criteria:

* History of Glaucoma
* History of hearth disease
* History of Alzheimer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
High intraorbital pressure | 1 minute
  IOP 18-22 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Ozhan Caparlar, Study Director — University of Health Dıskapı Yıldırım Beyazıt Training and Hospital
Locations (1):
- University of Health Dıskapı Yıldırım Beyazıt Training and Hospital, Ankara, Altındag, Turkey (Türkiye)

REFERENCES:
- [Background] Griesdale DE, Liu D, McKinney J, Choi PT. Glidescope(R) video-laryngoscopy versus direct laryngoscopy for endotracheal intubation: a systematic review and meta-analysis. Can J Anaesth. 2012 Jan;59(1):41-52. doi: 10.1007/s12630-011-9620-5. Epub 2011 Nov 1. PMID 22042705
- [Result] Vinayagam S, Dhanger S, Tilak P, Gnanasekar R. C-MAC(R) video laryngoscope with D-BLADE and Frova introducer for awake intubation in a patient with parapharyngeal mass. Saudi J Anaesth. 2016 Oct-Dec;10(4):471-473. doi: 10.4103/1658-354X.179118. PMID 27833500